CLINICAL TRIAL: NCT07083856
Title: Comparison of the Effects of Reiki and Self-Acupressure Applications on Functionality and Quality of Life in Patients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Effects of Reiki and Self-Acupressure Applications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, PhD, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/ 11- 14
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Reiki; Self-Acupressure; Functionality; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The groups doing the analysis will do the analysis without knowing it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki group (Experimental): Group where Reiki was applied
  Interventions: Behavioral: Reiki
- Self-acupressure applied group (Experimental): Group where Self-acupressure was applied
  Interventions: Behavioral: Self-Acupressure
- Control (No Intervention): Group with no intervention

INTERVENTIONS:
Behavioral: Reiki — Reiki
  Arms: Reiki group
Behavioral: Self-Acupressure — Self-Acupressure
  Arms: Self-acupressure applied group

SUMMARY:
Reiki, the subject of our research, is a complementary medicine practice within energy approaches. Discovered in Sanskrit texts by Dr. Usui in Japan in the late 19th century, it was demonstrated through studies demonstrating its effectiveness in symptoms of pain, depression, insomnia, and fatigue. Everything in the universe, including the human body, is composed of energy; any disruption in this energy can lead to illness. There are seven chakras where Reiki is applied. The main chakra centers are located along the spine. During Reiki treatments, the hands are held in each position, touching the head, neck, chest, abdominal cavity, and groin for 3-5 minutes. This period may extend to 10-20 minutes in problematic areas. The average treatment duration is 30-90 minutes. During the treatment, the patient lies down or reclines, and there is no need to remove clothing. During Reiki treatment, individuals may report a slight warming sensation under or near the therapist's hand. The only rule in Reiki practice is that the individual gives the practitioner permission to facilitate the flow of energy. The person receiving Reiki does not need to believe in Reiki during the treatment. Reiki is a universal life energy present in everyone. Reiki is generally safe, and no serious side effects have been reported. Over the last 10 years, Reiki practice has been increasing among physicians, nurses, and other healthcare professionals. This study will compare the effects of acupressure and Reiki treatments on functionality and quality of life in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to participate
2. Patients who have no communication problems
3. Patients who are 18 years of age or older
4. Patients who live in the center
5. Patients who have no scratches or deformities in the treatment area
6. Patients who do not smoke, use drugs, or use tranquilizers, and are not pregnant
7. Patients who have been receiving MS treatment for more than three months

Exclusion Criteria:

1. Patients who smoke, use substances, or use tranquilizers
2. Have dyspnea
3. Have anemia
4. Have diabetes
5. Have received corticosteroid treatment in the last three months
6. Have had an MS attack in the last three months
7. Have an autoimmune disease other than multiple sclerosis
8. Have signs of infection
9. Have a thyroid problem
10. Are taking psychostimulant medications
11. Have anxiety or depression detected in outpatient clinic screenings
12. Refuse to participate in the study
13. Have another known neurological system disease (dementia, Alzheimer's, etc.)
14. Have a communication barrier will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
The Multiple Sclerosis Quality of Life | 4 weeks
  The Turkish adaptation of the scale was conducted by Tülek in 2006. Tülek found Cronbach's alpha reliability coefficients to be 0.94 for the composite physical health and 0.89 for the composite mental health. This scale was created by adding 18 items related to MS-specific problems to the items related to general health perception (5 items), energy/fatigue (5 items), social functioning (2 items), emotional well-being (5 items), role limitations due to emotional problems (3 items), physical functioning (10 functions), role limitations due to physical problems (4 items), pain (3 items), and health changes found in the SF-36, a widely used generic quality of life scale for many conditions. The MSQOL-54 Quality of Life Scale consists of two main groups: physical health composite and mental health composite, 13 subgroups, and two independent items. Scores range from 0 to 100, with higher scores indicating higher quality of life.
The Multiple Sclerosis Functional Composite | 4 weeks
  The Scale consists of three subtests: the "9-Hole Peg Test" that evaluates upper extremity functions, the "25-Step Walking Test" that checks lower extremity functions, and the "Step Auditory Serial Addition Test" that evaluates immediate memory and cognitive functions. It was administered within the MSFC.

CONTACTS AND LOCATIONS:
Overall Officials: Caner F Demir, MD, Study Chair — Firat University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Fethi̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No